CLINICAL TRIAL: NCT04651608
Title: Effectiveness of Acupress in The Management of Chemotherapy-Developed Acute Nausea Vomiting Symptoms In Child Oncology Patients
Brief Title: The Effect of Acupressure Chemotherapy-related Nausea Vomiting in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Duygu ALTUNTAŞ BALCI, lecturer, Akdeniz University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TYL-2016-1099; TYL-2016-1099 (Other: Akdeniz Üniversitesi)
Record Dates: First submitted 2020-07-21; First posted 2020-12-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Pediatric Cancer; Nausea With Vomiting Chemotherapy-Induced
Keywords: nursing; child cancer patients; acupressure; Nausea with Vomiting Chemotherapy-Induced; nausea and vomiting; pediatric cancer
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: One of the 2 procedure groups randomized with sealed envelope was applied acupressure with pressure to the P-6 point on the wrist of the child by the researcher in the first application, the other is applied with sea-band, and it was followed for 24 hours. Acupressure application was performed on both wrists for 2 minutes each with pressure, and 15 minutes each with sea-band. In the next chemotherapy treatment, a placebo of the first procedure (placebo pressure/placebo sea-band) was applied to each child, which ensured the control group of their own.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manuel acupressure (Experimental): In this group, manual acupress was applied to children receiving chemotherapy with moderate and high emetogenic effects.
  Interventions: Behavioral: manuel acupressure; Behavioral: placebo manuel acupressure
- sea-band acupressure (Experimental): In this group, sea-band acupressure was applied to children receiving chemotherapy with moderate and high emetogenic effects.
  Interventions: Behavioral: sea-band acupressure; Behavioral: placebo sea-band

INTERVENTIONS:
Behavioral: manuel acupressure — Acupressure was applied once by the researcher 30 minutes before applying the chemotherapeutic agent with medium or high emetogenicity to the randomized child. 3 fingers were placed on the child's wrist with their fingers and the region (point P6) between the flexor carpi radians and palmaris longus 1 cm below. Acupressure was applied to the wrist of the child by press for 2 minutes. The same procedure was applied to the other wrist. Then, data were recorded in accordance with the data collection procedure.
  Arms: manuel acupressure
Behavioral: sea-band acupressure — 30 minutes before applying the chemotherapeutic agent with medium or high emetogenicity to the randomized child, sea-band acupress was applied by the researcher. The P6 point on the wrist was identified and marked with the child's own fingers. A sea band was attached to both wrists of the child by the researcher. The attached sea-band was allowed to remain for 15 minutes and was removed by the researcher at the end of the period. Separate sea-band was attached to each child. Acupress wrist bands, which are produced in separate sizes for adults and children, were used during the application, taking into account the physical development of the child, pediatric for the age range of 5-12, and adult size sea-band for the age of 12. Acupress application with sea-band was done once. Then, data were recorded in accordance with the data collection procedure
  Arms: sea-band acupressure
Behavioral: placebo manuel acupressure — Placebo manual acupress was applied in the next protocol for the child who was administered manual acupressure.
  Arms: manuel acupressure
Behavioral: placebo sea-band — Placebo sea-band was applied in the next protocol for the child who was administered sea-band acupressure.
  Arms: sea-band acupressure

SUMMARY:
This study is carried out to evaluate and compare the efficiency of acupressure practice applied with pressure or sea-band and their placebo on managing the acute nausea-vomiting symptoms developing due to chemotherapy in pediatric oncology patients.

DETAILED DESCRIPTION:
Every year children aged 0 to 19 years old are diagnosed with cancer around the world. For pediatric oncology patients, chemotherapy-related acute nausea and vomiting are among most common symptoms and has a bad influence on quality of life. When it cannot be prevented, it can cause serious medical problems. Continuous, repetitive and unavoidable vomiting affects patients' and their families' quality of life adversely, causing delay or even termination in chemotherapy treatment. It is a well-known fact that medical treatment is insufficient to control nausea and vomiting symptoms. Therefore, supportive care is needed besides medical treatment. One of the approaches mentioned is acupressure. Non-invasive stimulation of the P6 acupuncture point is a harmless and complementary approach to health. The point between flexor carpi radialis and palmaris longus, located at a three finger distance from the wrist crease, is named as "P6 Nei-Guan". This acupuncture point, placed on the pericardium channel, is generally used to harmonize stomach and relieve the vomiting. Acupressure is a way of stimulation applied on acupuncture points by finger, palm or acustimulation bands (sea-band, relief band) and can be used for children as well. Acupressure is defined as one of the complementary health approaches which nurses can apply. It is stated that this method, which is non-invasive, economical, easy to apply and reliable, has no side effect and patients can apply to themselves with a good guidance.

Chemotherapy-related nausea and vomiting are among the symptoms affecting children's quality of life and their adaptation to the treatment. There are limited amount of research intended to manage pediatric oncology patients' chemotherapy-related nausea and vomiting symptoms by using acupressure. It is thought that the research will provide significant contribution for literature, nursing practice and the quality of patient care since power of the study is high and it is the first study which efficiency of wrist-band, manuel acupressure and placebos is being compared for management of chemotherapy-related acute nausea and vomiting symptoms in pediatric oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 5-18,
* Who have a chemotherapy protocol with a high and moderate emetogenic effect according to MASCC / ESMO Antiemetic Guidance Classification
* Not having a verbal communication disorder.

Exclusion Criteria:

* If the participants did not receive chemotherapy or were receiving it for the first time,
* Branching, redness, phlebitis, edema, open wound, fracture, infection, etc. in the wrist
* Any obstacles for the verbal assessment of the child (intubation, etc.).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
number and severity of nausea, number and severity of vomiting | during study
  Following the interventions, the number of nausea and vomiting experienced by children was followed up for 24 hours. visual severity scale was used to score nausea and vomiting severity. (numeric expression, VAS, 0-10)

SECONDARY OUTCOMES:
antiemetic need | during study
  The antiemetic drugs needed by children were recorded for 24 hours after the interventions. (numeric expression, 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Aysegül İŞLER DALGIÇ, Professor, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data sharing plans for the current study are unknown and will be made available at a later date.

REFERENCES:
- [Background] Dupuis LL, Kelly KM, Krischer JP, Langevin AM, Tamura RN, Xu P, Chen L, Kolb EA, Ullrich NJ, Sahler OJZ, Hendershot E, Stratton A, Sung L, McLean TW. Acupressure bands do not improve chemotherapy-induced nausea control in pediatric patients receiving highly emetogenic chemotherapy: A single-blinded, randomized controlled trial. Cancer. 2018 Mar 15;124(6):1188-1196. doi: 10.1002/cncr.31198. Epub 2017 Dec 19. PMID 29266260
- [Background] Jones E, Isom S, Kemper KJ, McLean TW. Acupressure for chemotherapy-associated nausea and vomiting in children. J Soc Integr Oncol. 2008 Fall;6(4):141-5. PMID 19134445
- [Background] Miao J, Liu X, Wu C, Kong H, Xie W, Liu K. Effects of acupressure on chemotherapy-induced nausea and vomiting-a systematic review with meta-analyses and trial sequential analysis of randomized controlled trials. Int J Nurs Stud. 2017 May;70:27-37. doi: 10.1016/j.ijnurstu.2017.02.014. Epub 2017 Feb 14. PMID 28231440